CLINICAL TRIAL: NCT06412237
Title: An Exploratory Study of a Wearable Robotic Hand Orthosis in the Chronic Stroke Population in Singapore: A Clinic to Home Feasibility Trial
Brief Title: An Exploratory Study of a Wearable Robotic Hand Orthosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB2023/00448
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Hand exoskeleton robot; Robotic hand orthosis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single site, pilot, feasibility study that focuses on the transition of technology use from the clinic to home environment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RELab tenoexo (Experimental): 3 weeks in clinic training (9 training sessions, two clinical assessment and 2 usability evaluations) followed by 2 weeks home training (1-hour daily training and to the extent participants desire). Lastly 1-month follow up clinical assessment and IMU data collection.
  Interventions: Device: RELab tenoexo

INTERVENTIONS:
Device: RELab tenoexo — The RELab tenoexo is a fully wearable and portable RHO developed at the Rehabilitation Engineering Laboratory (RELab) at ETH Zurich.

SUMMARY:
Upper limb deficits usually remain in 75% of the stroke survivors despite completing full rehabilitation. This is due to lack of effectiveness of rehabilitation and the degree of support and resources available.

In this study, the investigators plan to study the use of assistive technologies in chronic stroke survivors.

DETAILED DESCRIPTION:
Assistive technologies have shown promising results in immediate improvement in functional abilities.

RELab tenoexo is a fully wearable and portable robotic hand orthoses (RHO) used for functional training. Its design support end users with functional hand opening and closing and can be applied in therapy exercises or during functional activities. While prior research demonstrated its effectiveness for spinal cord injury, it hasn't been tailored for multi-ethnic stroke populations.

This study aims to determine the feasibility and extent to which the RELab tenoexo can complement therapy training in clinic and further be used as both a training and assistive device in the home environment. In addition, it also aims to investigate the amount of upper limb usage before, during and after the training period.

ELIGIBILITY:
Inclusion Criteria:

* Patient with first ever clinical stroke (ischaemic or haemorrhagic) with hemiplegic motor deficit(s) due to stroke as diagnosed by CT or MRI.
* Post stroke of at least 6 months with stable neurological status.
* Age 21 to 80 years of age.
* Hemiplegic pattern and shoulder abduction MRC motor power > 2/5 and elbow extension >2/5
* Has a stable home abode and a carer/NOK to assist with donning of device and supervise home based exercise
* MOCA > or equal to 22/30
* Able to give and sign informed consent at research site.
* Able to speak English

Exclusion Criteria:

* Non-stroke related causes of arm motor impairment.
* Has unstable or terminal medical conditions which may affect participation (e.g.: unresolved sepsis, postural hypotension, end stage renal failure, cancer, retroviral disease, on immunosuppressive therapy) or anticipated life expectancy of <1 year due to malignancy or neurodegenerative disorder.
* Local factors which may be worsened by intensive arm therapy: spasticity of Modified Ashworth Scale grades 3-4, skin wounds, shoulder pain Pain Scale >5/10, active/non-united fractures or arthritis or fixed joint/tissue flexion contractures of shoulder, elbow, wrist or fingers incompatible with tenoexo interface.
* Patient with severe cognitive, perceptual (include hemi-neglect), and/or emotional-behavioural issues that preclude participation.
* Experiencing moderate to severe levels of pain (Numerical Vertical Pain Scale > 5).
* Is pregnant or breast feeding. Neither the tenoexo nor the IMUs have been tested to evaluate the usage with pregnant and/or breast feeding mothers. Further, due to the length of the study, pregnancy may make it difficult to follow the study schedule.
* Have a pacemaker. Magnets are used throughout the system.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) Score | Week 2 (baseline), 4 (end of in-clinic training) ,8 (end of home training) ,12 (follow-up assessment)
  Functional and dexterity score in the affected arm evaluated using 19 tests of motor function across 4 subsets; minimum score = 0, maximum score = 57, with higher score indicating better function.

SECONDARY OUTCOMES:
Fugl-Meyer Motor Assessment (FMA) scale | Week 2 (baseline), 4 (end of in-clinic training) ,8 (end of home training) ,12 (follow-up assessment)
  Change in Fugl Meyer Motor Assessment score in the affected arm, minimum: 0, maximum: 66 with higher scores indicating greater levels of mobility function
Grip Strength (kg) | Week 2 (baseline), 4 (end of in-clinic training) ,8 (end of home training) ,12 (follow-up assessment)
  Measured by Digital hand-held Dynamometer (mean of 3 readings) for both hands
Hr-QOL scales using SS-QOL (Stroke specific Quality of Life scale) | Week 2 (baseline), 4 (end of in-clinic training) ,8 (end of home training) ,12 (follow-up assessment)
  Quality of life scale specific to stroke patients, minimum 49, maximum 245; with higher scores indicating better function.
EQ-5D-5L scale | Week 2 (baseline), 4 (end of in-clinic training) ,8 (end of home training) ,12 (follow-up assessment)
  Standardized measure of health-related quality of life using a 5 level scale (no problem, slight problems, moderate problems, severe problems, unable to)
Self-efficacy outcomes by UPSET (upper limb self-efficacy test) | Week 2 (baseline), 4 (end of in-clinic training) ,8 (end of home training) ,12 (follow-up assessment)
  Questionnaire to measure self-efficacy in various tasks after stroke
System Usability Scale (SUS) | Week 3 (mid in-clinic training), 4 (end of in-clinic training), 8 (end of home training)
  To assess the overall usability of the tenoexo (effectiveness, efficiency, satisfaction), scaled from 1 (Strongly disagree) to 5 (Strongly Agree)
Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) | Week 3 (mid in-clinic training), 4 (end of in-clinic training), 8 (end of home training)
  To evaluate user satisfaction with assistive technology, scaled from 1 (Not satisfied at all) to 5 (Very satisfied)

OTHER OUTCOMES:
Modified Ashworth Scale (MAS) | Week 2 (baseline), 4 (end of in-clinic training) ,8 (end of home training) ,12 (follow-up assessment)
  Measures the level of spasticity at the elbow and finger flexors of proximal interphalangeal joint regions; scored from "0 to 4" with "4" indicating affected part is more spastic in flexion/extension.
Visual Analogue Scale (self-reported pain score) | Week 2 (baseline), 4 (end of in-clinic training) ,8 (end of home training) ,12 (follow-up assessment)
  Unidimensional measure of pain intensity; "0" being no pain and "10" being worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Tegan Plunkett, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanczak N, Plunkett TK, Lin S, Kuenzler L, Lau M, Kuah WKC, Ng CY, Gassert R, Chua K, Lambercy O. Feasibility of post-stroke hand rehabilitation supported by a soft robotic hand orthosis in-clinic and at-home. J Neuroeng Rehabil. 2025 Aug 21;22(1):183. doi: 10.1186/s12984-025-01717-6. PMID 40842028